CLINICAL TRIAL: NCT06426576
Title: Application of Load Limits After Orthopaedic Surgery With Biofeedback-based Instructions Compared to a Conventional Method
Brief Title: Load Limits After Orthopaedic Surgery: Biofeedback vs. Conventional Method (AppPWB)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-00106; mu24Mauch
Record Dates: First submitted 2024-05-17; First posted 2024-05-23 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Surgery
Keywords: Orthopaedic surgery; Partial weight bearing; Portable measurement systems; Plantar pressure insoles; Biofeedback function

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): The control group receives instructions on partial weight bearing using the standard method.
  Interventions: Other: Standard one-off instruction using a scale
- Intervention group (Experimental): The intervention group receives instructions on partial weight bearing using a plantar pressure sole inserted into the shoe that measures the force/weight applied to the foot and indicates the applied weight to the patient both visually and acoustically via a smartphone app.
  Interventions: Device: Plantar pressure insoles

INTERVENTIONS:
Other: Standard one-off instruction using a scale — The permitted weight is demonstrated to the patient once using a scale in the static position. The patient repeatedly places the foot with the permitted weight on a scale in order to develop a feeling for the load. After this exercise in the static position, the patient applies the perceived load to dynamic activities of daily living without receiving any feedback.
  The instruction is given by a trained physiotherapist. Simultaneously with the instruction, the effective weight applied on the leg will be measured using instrumented insoles without any feedback.
  Arms: Control group
Device: Plantar pressure insoles — The insoles are used in both static and dynamic conditions such as walking straight along the hallway or walking stairs if applicable. Initial instruction is given by a trained physiotherapist and will be continuously applied at home using the smartphone app for 5 out of 7 days per week during the first 2 weeks after surgery.
  Arms: Intervention group

SUMMARY:
The aim of this single-centre prospective randomized-controlled clinical trial is to assess whether patients adhere to prescribed weight bearing limits after surgical orthopaedic or traumatological interventions more accurately after instruction using a biofeedback method than using the standard method.

DETAILED DESCRIPTION:
Partial weight bearing, commonly prescribed post-surgery in orthopaedics and traumatology, aims to stimulate healing while preventing overloading. Partial weight bearing refers to that the patient is only allowed to put 10 to 50% of their body weight on the affected limb.

The most commonly used method for instructing partial weight bearing with the patient is using a personal scale. This means that the patient can only exercise in a static position and the perceived load must be transferred to dynamic activities of daily living without further feedback. Previous reports indicate that patients often struggle to adhere to prescribed partial weight-bearing limits, frequently exceeding the specified load by 100% or more. However, when additional feedback was incorporated into training, approximately 90% of subjects successfully adhered to the partial load.

Portable or wearable measuring systems, such as pressure-sensitive insoles, offer feedback during dynamic tasks, facilitating a smoother transition to daily activities. Unlike the standard one-time instruction using a scale, these systems provide repeated feedback at each step, promoting a higher frequency of exercises. This aids patients in developing a better sense of the correct load.

This single-centre prospective randomized-controlled clinical trial aims to investigate the effectiveness of pressure insoles connected to a smartphone via Bluetooth and operated using an app in improving partial weight bearing adherence. The insoles provide direct feedback through acoustic and visual signals if the affected leg is overloaded, possibly leading to a lower proportion of steps over the load limit compared to those without feedback. Participants are randomized into either the intervention group (dynamic condition - plantar pressure insoles) or the control group (static condition - standard one-off instruction using a scale).

The primary objective is to determine whether the proportion of steps exceeding the weight bearing limit is lower in the intervention group compared to the control group 2 weeks after surgery. Secondary objectives include assessing subjective ratings of the permitted load, perceived pain, and mobility. Additionally, the trial hypothesizes that patients using the insoles can estimate applied load more accurately. The intervention group will also provide feedback on the usability of the app and insoles.

The results of this trial will contribute to enhancing postoperative treatment of patients undergoing orthopaedic surgery, thereby improving treatment outcomes and optimizing therapy regimens.

ELIGIBILITY:
Inclusion Criteria:

* Patients with prescribed partial weight bearing (joint-independent) for at least 2 weeks
* Unilateral injury of the lower extremity
* Having their own smartphone
* Age 18 years and older

Exclusion Criteria:

* Patients with prescribed full weight bearing
* Patients with prescribed complete unloading
* Patients with prescribed self-selected loading "according to pain"
* Bilateral injuries of lower extremities
* Upper extremity injuries precluding the use of crutches
* Use of walking aids prior to injury
* Neurological conditions affecting gait
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc.,
* Previous enrolment in a clinical trial
* Body mass > 135 kg
* Age under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Proportion of steps (%) over of the prescribed weight bearing limit on the injured leg while walking, assessed with the instrumented insoles. | At 2 weeks post-surgery
  After 2 weeks of continuous use of the feedback-providing insoles by the intervention group, the adherence to load limits is evaluated at the follow-up visit. This assessment aims to determine if the intervention group adheres better to the prescribed weight-bearing limits compared to the control group, which did not receive feedback during this period. Both groups have the proportion of steps (%) exceeding the prescribed weight-bearing limit on the injured leg while walking assessed using instrumented insoles.

SECONDARY OUTCOMES:
Assessment of perceived pain | Baseline and at 2 weeks post-surgery
  To assess the pain level, the numeric analog scale is used. Patients are asked to rate their pain on a scale from 0 to 10, where 0 indicates no pain while 10 indicates the worst possible pain.
Assessment of physical activity | Baseline and at 2 weeks post-surgery
  To assess the physical activity, the UCLA Activity Scale(UCLA) is used The UCLA Activity Scale consists of questions related to different activities, and patients rate their ability to perform each activity on a scale from 1 to 10, with higher scores indicating greater activity levels.
Assessment of mobility | Baseline and at 2 weeks post-surgery
  To assess the mobility, the Life Space Questionnaire and Parker Mobility Score are used. The former asks respondents to report on their frequency of movement and the distance traveled within various zones, such as within their home, neighborhood, and beyond. The latter evaluates an individual's ability to perform three basic mobility tasks. A score is given to each activity on a 4 point scale (0 - not at all, 1 - assistance of one person, 2 - with an aid, 3 - no difficulty and no aid) and then combined to provide a final score between 0 and 9, where 9 is independent with no aid in all three activities, and 0 is not able to carry out any of the activities.
Assessment of the quality of life | Baseline and at 2 weeks post-surgery
  The health-related quality of life is assessed using the EuroQol-5 Dimensions (EQ-5D). It is a standardized questionnaire used to assess an individual's health status across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has three levels of severity (no problems, some problems, extreme problems), allowing for the classification of 243 unique health states.
Assessment of perceived load applied | At 2 weeks post-surgery
  Patients are asked to estimate the applied load.
Assessment of the usability of the planar pressure insoles (intervention group only) | At 2 weeks post-surgery
  The intervention group is asked to provide feedback on the usability of the app and insoles using a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Marlene Mauch, Dr., Principal Investigator — Department of Orthopaedics and Traumatology, University Hospital Basel
Locations (1):
- Department of Orthopaedics and Traumatology, University Hospital Basel, Bethesda Spital Basel, Basel, Canton of Basel-City, Switzerland